CLINICAL TRIAL: NCT07363863
Title: Pattern of Treatment and Outcomes of Locally Advanced Rectal Carcinoma : a Retrospective Study
Brief Title: Pattern of Treatment and Outcomes of Locally Advanced Rectal Carcinoma
Status: Not yet recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Azhar Abdelgaber Moez Abdelraheem, principal investigator, Sohag University
Other Study IDs: Soh-Med--25-11-2MS
Record Dates: First submitted 2025-11-27; First posted 2026-01-23 (Actual); Last update posted 2026-01-23 (Actual); Status verified 2025-11

CONDITIONS: Rectal Carcinoma
MeSH Terms: conditions — Rectal Neoplasms | interventions — saxagliptin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: No Intervention (subjects were previously treated with Onglyza®) — no intervention

SUMMARY:
the study will discuss different pattern of treatment and the outcomes of locally advanced rectal carcinoma as a retrospective study.

The study will be conducted at Department of Clinical Oncology, Sohag University Hospital and Sohag Cancer center, Sohag, Egypt.

including patients diagnosed and treated between 2018 and 2025. and the data will be collected from reports .

ELIGIBILITY:
Inclusion Criteria:

* patients who were more than18 years old at time of diagnosis.
* Patients with histologically confirmed rectal carcinoma.
* Stage II-III (locally advanced) disease at initial diagnosis.

Exclusion Criteria:

* Patients with distant metastasis at presentation.
* Patients diagnosed with double malignancy.
* Patients with incomplete medical records.
* Organ failure

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study will be conducted at Department of Clinical Oncology, Sohag University Hospital and Sohag Cancer center, Sohag, Egypt.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-10-01 (Estimated)

PRIMARY OUTCOMES:
Estimation of overall survival (OS ). | 2018 _ 2025
Estimation of Response rate . | 2018-2025
Estimation of disease-free survival (DFS) . | 2018-2025

SECONDARY OUTCOMES:
treatment-related toxicity: (graded by CTCAE v5). | 2018-2025